CLINICAL TRIAL: NCT02173093
Title: Treatment of Neuroblastoma and GD2-Positive Tumors With Activated T Cells Armed With OKT3 X Humanized 3F8 Bispecific Antibodies (GD2Bi): A Phase I/II Study
Brief Title: Activated T Cells Armed With GD2 Bispecific Antibody in Children and Young Adults With Neuroblastoma and Osteosarcoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Daniel W. Lee, MD, Principal Investigator, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19031; NCI-2014-01149 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2013-171 (Other: Barbara Ann Karmanos Cancer Institute); P30CA022453 (NIH)
Record Dates: First submitted 2014-06-22; First posted 2014-06-24 (Estimated); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Disseminated Neuroblastoma; Recurrent Neuroblastoma
Keywords: Neuroblastoma; Solid tumor; Immunotherapy targeting GD2; Bispecific antibodies; Activated T cells
MeSH Terms: conditions — Neuroblastoma | interventions — Interleukin-2; aldesleukin; Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (IL-2, GM-CSF, GD2Bi-aATC) (Experimental): Patients receive IL-2 SC daily on days -2 to 35, GM-CSF SC twice weekly x 5 weeks, and GD2Bi-aATC IV over 30 minutes twice weekly x 4 weeks for a total of 8 infusions. Laboratory evaluations of immune responses are obtained prior and after immunotherapy.
  Interventions: Biological: IL-2; Biological: GD2Bi-aATC; Biological: GM-CSF; Other: laboratory evaluations of immune responses

INTERVENTIONS:
Biological: IL-2 — Given SC
  Other Names: aldesleukin; Proleukin; recombinant human interleukin-2; recombinant interleukin-2
Biological: GD2Bi-aATC — Given IV
  Other Names: GD2Bi-armed aATC
Biological: GM-CSF — Given SC
  Other Names: sargramostin; Leukine; Prokine
Other: laboratory evaluations of immune responses — Correlative studies
  Other Names: laboratory biomarker analysis

SUMMARY:
Previous research has demonstrated that investigators can coat (arm) T cells with a special molecule called GD2 bispecific antibody that will help T cells recognize neuroblastoma and osteosarcoma cells and kill them. This bispecific antibody recognizes GD2, a protein found on almost all neuroblastoma and osteosarcoma cells. The investigators put the GD2 bispecific antibody on T cells and give large numbers of these T cells back to patients. The investigators think that these T cells may have a better chance of killing GD2 expressing tumor cells when they are armed with GD2 bispecific antibody. This trial studies the side effects and best dose of activated T cells armed with GD2 bispecific antibody and how well they work in treating patients with neuroblastoma, osteosarcoma, and other GD2-positive solid tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To perform a phase I dose-escalation study in patients with recurrent or refractory neuroblastoma (NB) and other GD2-positive tumors to evaluate the safety and tolerability and to determine the maximum tolerated dose (MTD) for anti-CD3 x hu3F8 bispecific antibody (GD2Bi)-armed activated T cells (aATC) infused twice a week for a total of eight infusions in combination with daily IL-2 (300,000 IU/m^2/day) and GM-CSF (250 ug/m^2 twice per week) in a standard 3 + 3 dose escalation schema with 40, 80, and 160 x 10^6 cells/kg/infusion dose levels.

II. To conduct a phase II clinical trial to explore efficacy and confirm the toxicity profile of GD2Bi-aATC combined with IL-2 and GM-CSF in a phase II expansion cohort of 22 patients with neuroblastoma (NB) using MTD determined in the phase I.

SECONDARY OBJECTIVES:

I. Evaluate immune responses in the phase I/II trial by sequential monitoring of anti-NB cytotoxicity of peripheral blood lymphocytes and IFN-gamma EliSpots directed at NB lines.

II. To evaluate persistence of aATC in the blood and tumor biopsies by staining for murine IgG2a to confirm trafficking of armed T cells to tumor.

III. To conduct exploratory study of (18F FDG) positron emission tomography (PET)/computed tomography (CT) after armed ATC infusions in selected patients with PET/CT measurable soft tissue and skeletal lesions.

OUTLINE: This is a phase I, dose-escalation study of OKT3/humanized 3F8 bispecific antibody-aATC followed by a phase II study.

Patients receive IL-2 subcutaneously (SC) daily on days -2 to 35, sargramostim SC twice weekly for 4 weeks, and OKT3/humanized 3F8 bispecific antibody-aATC intravenously (IV) over 30 minutes twice weekly for 4 weeks.

After completion of study treatment, patients are followed up at 1, 3, 6, and 12 months.

ELIGIBILITY:
The study is now in the phase II expansion phase.

Inclusion Criteria for phase II:

* The target tumor is limited to neuroblastoma and the diagnosis should be histologically verified.
* Patients must have refractory or recurrent malignancy; patient's current disease state must be one for which no known curative therapy is available;
* Patients should not receive any other experimental or phase 1 therapy within 3 weeks prior to study enrollment and monoclonal antibody therapy within 6 weeks
* To be eligible for phase I study patients should have primary refractory or relapsed disease as evidenced by:

  * Local tumor recurrence measurable on CT or magnetic resonance imaging (MRI) scans with or without metastatic lesions
  * Refractory bone marrow involvement in patients with NB
  * NB with MIBG-positive skeletal lesions
* The presence of radiographically measurable disease immediately prior to start of Phase I immunotherapy is not an eligibility requirement in the following situations:

  * In patients with NB who have documented bone marrow (BM) involvement;
  * In patients with NB who have MIBG-positive bony lesion(s);
* An additional eligibility requirement for phase II study includes the presence of radiographically measurable disease with the exception of MIBG-positive NB or NB with bone marrow involvement:
* Patients must have a Lansky or Karnofsky performance status score of >= 70
* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy

  * Myelosuppressive chemotherapy: must not have received within 3 weeks of starting immunotherapy (IT)
  * Hematopoietic growth factors: at least 7 days since the last dose of growth factor therapy
  * Immunotherapy: at least 6 weeks must have elapsed since prior therapy that includes a monoclonal antibody
* Normal organ function
* All patients or their parents or legal guardians must sign a written informed consent; assent, when appropriate, will be obtained according to institutional guidelines
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Exclusion Criteria:

* Patients who are pregnant or breast-feeding are not eligible for this study; negative pregnancy tests must be obtained in girls who are postmenarchal; males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method for the duration of study therapy and for 3 months after the last dose of GD2Bi-aATC; breastfeeding women should be excluded
* Patients who have an uncontrolled infection are not eligible
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible

Ages: 13 Months to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-11; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of GD2Bi-aATC | 35 days
  Safety of GD2Bi-aATC infusions is evaluated to determine MTD

SECONDARY OUTCOMES:
Anti-tumor activity | Up to 12 months
  Objective response rate to GD2Bi-aATC infusions
Immune responses after GD2Bi-aATC infusions | Up to 12 months
  In vitro anti-tumor activity of patients' lymphocytes; changes in cytokine profile; changes in lymphocyte phenotypes

CONTACTS AND LOCATIONS:
Overall Officials: Maxim Yankelevich, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (3):
- United States (3):
  - Children's Hospital of Michigan, Detroit, Michigan
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Virginia, Department of Pediatrics, Hematology/Oncology, Charlottesville, Virginia

REFERENCES:
- [Derived] Park JA, Santich BH, Xu H, Lum LG, Cheung NV. Potent ex vivo armed T cells using recombinant bispecific antibodies for adoptive immunotherapy with reduced cytokine release. J Immunother Cancer. 2021 May;9(5):e002222. doi: 10.1136/jitc-2020-002222. PMID 33986124